CLINICAL TRIAL: NCT03527017
Title: Cross-Sectional Survey on the Use of Tobacco Products in the General Population and in Users of IQOS in Germany (2018-2020)
Brief Title: Cross-Sectional Survey on the Use of Tobacco Products - Germany
Status: Terminated | Type: Observational
Why Stopped: The study was terminated prematurely after 2 years because during to the COVID-19 pandemic, the face-to-face mode of administration of the interviews in the General Adult Population Sample was not feasible.
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: P1-PMX-03-DE
Record Dates: First submitted 2018-05-04; First posted 2018-05-16 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Tobacco Use
Keywords: Tobacco Use; IQOS
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General Population: Adults living in Germany.
  Interventions: Other: Survey on Use of Tobacco Products in the General Population
- IQOS Users: Adult current IQOS users (at the time of survey) living in Germany who are registered in the Germany IQOS User Database and agreed to be contacted for research purposes at the time of registration.
  Interventions: Other: Survey on Use of Tobacco Products in IQOS Users

INTERVENTIONS:
Other: Survey on Use of Tobacco Products in the General Population — Face-to-face survey to estimate the prevalence of current tobacco use status in the general population of Germany.
  Groups: General Population
Other: Survey on Use of Tobacco Products in IQOS Users — Online survey to describe patterns of use in adult IQOS users residing in Germany.
  Groups: IQOS Users

SUMMARY:
The main purpose of the research study is to estimate the prevalence of tobacco product use and describe the tobacco use patterns in adults in Germany.

DETAILED DESCRIPTION:
The aim of the survey is to describe the current and past patterns of use of tobacco products in the general adult population of Germany and in adult IQOS users registered in the IQOS user database of Philip Morris GmbH (Germany IQOS User Database), and explore their association with key independent variables. More specifically, the objectives are:

1. Estimate the prevalence of current tobacco use status in the study population.
2. Describe the past tobacco use status (cigarette, IQOS and other innovative products, including e-cigarettes) in the study population (i.e. never-use, initiation, product use transition, cessation, re-initiation, and relapse).
3. Explore the association between self-reported health status and use of tobacco products in the study population.
4. Explore the association between patterns of use (including misuse) with motivation to use, perceived quality attributes of IQOS (e.g. risk and self-reported changes since switching to the product, in a number of relevant domains where IQOS may have potential benefits), and consumer's satisfaction in the population of IQOS users in Germany registered in the Germany IQOS User Database.

ELIGIBILITY:
Inclusion Criteria (all participants, including IQOS users):

* Legally permitted to buy tobacco products in Germany (≥18 years of age).
* Currently residing in Germany.
* Able to read, write and understand German.
* Consent to participate in the survey

Inclusion Criteria (IQOS users only):

* Has used more than 100 HEETS tobacco sticks in his or her lifetime.
* Is currently using IQOS.
* Has access to the internet.
* Is not currently employed by Philip Morris International or any of its affiliates

Exclusion Criteria:

* Not meeting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be limited to residents of Germany.
Sampling Method: Probability Sample
Enrollment: 6284 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Prevalence of current tobacco use | Study duration (3 years).
  Prevalence of current tobacco use status in the study population.
Past tobacco use status | Study duration (3 years).
  Past tobacco use status (cigarette, IQOS and other innovative products) in the study population.
Self-reported health status | Study duration (3 years).
  Association between self-reported health status and use of tobacco products in the study population.
Perceived risk | Study duration (3 years).
  Association between patterns of use with perceived risk.
IQOS use experience | Study duration (3 years).
  Describe the IQOS user experience, including motivation to use, mis-use, satisfaction, and self-reported changes since switching to the product (in a number of domains where IQOS may have potential benefits).

CONTACTS AND LOCATIONS:
Overall Officials: Pierpaolo Magnani, Study Chair — Philip Morris Products S.A.
Locations (1):
- Philip Morris Products S.A., Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No